CLINICAL TRIAL: NCT03996460
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Impact of K0706 on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics and Clinical Outcomes in Dementia With Lewy Bodies (DLB)
Brief Title: K0706 for Patients Diagnosed With Dementia With Lewy Bodies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Principal Investigator, Fernando Pagan MD, Associate Professor Of Neurology , Director of Movement Disorder Program, Medical Director of NPF COE at GUH , Fellowship Director, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000266
Record Dates: First submitted 2019-06-13; First posted 2019-06-24 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease

STUDY DESIGN:
Intervention Model Description: The effects of 192 mg powder of K0706 ( equivalent to 96 mg capsule of K0706) versus 384 mg powder of K0706 (equivalent to 192 mg capsule of K0706) versus matching placebo powder taken daily by mouth for 12 weeks, followed by a 4 week wash-out period in individuals diagnosed with DLB will be evaluated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized by a Biostatistician by an internet based randomization module into three groups. The researchers include : Primary investigator , Sub-Investigators ,Clinical Coordinators, Nurse Practitioners, and Clinical Research unit (CRU) staff.
  The investigators will be blinded to the dosage. Medications for any patient will be labeled by the CRU with a package medical identification number (Med. Id). A patient specific patient identification number (Pat. Id.) will be assigned to each patient. The investigator will have to note the Pat.Id on the designated medication package number after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo powder (Placebo Comparator): Forty five (45) participants will be recruited and randomized into 3 arms (1:1:1). Fifteen (15) patients in arm 1 (group 1) will receive the matching placebo powder orally once daily for 12 weeks (90 days).
  Interventions: Drug: Placebo
- 192 mg powder of K0706 (Active Comparator): Forty five (45) participants will be recruited and randomized into 3 arms (1:1:1) .Fifteen (15) patients in arm 2 (group 2) will receive the 192 mg powder of K0706 ( equivalent to 96 mg capsule of K0706) orally once daily for 12 weeks (90 days).
  Interventions: Drug: 192 mg powder of K0706
- 384 mg powder of K0706 (Active Comparator): Forty five (45) participants will be recruited and randomized into 3 arms (1:1:1) .Fifteen (15) patients in arm 3 (group 3) will receive the 384 mg powder of K0706 (equivalent to 192 mg capsule of K0706) orally once daily for 12 weeks(90 days).
  Interventions: Drug: 384 mg powder of K0706

INTERVENTIONS:
Drug: Placebo — Fifteen (15) patients in group 1 will receive the sachet of matching placebo ( equivalent to a capsule of placebo"sugar pill") orally daily for 12 weeks (90 days) without food.
  Arms: Placebo powder
Drug: 192 mg powder of K0706 — Fifteen (15) patients in group 2 will receive the sachet of 192 mg powder of K0706 ( equivalent to 96 mg capsule of K0706) orally for 12 weeks (90 days) without food.
  Arms: 192 mg powder of K0706
Drug: 384 mg powder of K0706 — Fifteen (15) patients in group 3 will receive the 384 mg powder of K0706 (equivalent to 192 capsule of K0706) orally daily for 12 weeks (90 days) without food.
  Arms: 384 mg powder of K0706

SUMMARY:
This study evaluates the safety and tolerability of treatment with K0706 in Dementia with Lewy Bodies (DLB).

The hypothesis is that K0706 will be safe and tolerable and that this drug will alter CSF and plasma biomarkers in DLB. Clinical assessments of cognitive, behavioral and motor functioning will also be evaluated. A total of 45 participants will be randomized 1:1:1 into 3 groups (n=15/per group) to be treated with sachet of 192 mg powder of K0706 ( equivalent to 96 mg capsule of K0706) or sachet of 384 mg powder of K0706 (equivalent to 192 capsule of K0706) or sachet of matching placebo ( equivalent to a capsule of placebo) for 12 weeks, followed by 4-week wash-out period.

DETAILED DESCRIPTION:
Dementia with Lewy Bodies (DLB) is an alpha-synucleinopathy and the second most common form of dementia in the elderly. DLB shares striking neuropathological and clinical similarities with both Parkinson's disease (PD) and Alzheimer's disease (AD). DLB and PD are characterized by death of dopaminergic (DA) neurons in the nigro-striatal system and formation of intra-neuronal alpha-synuclein inclusions known as Lewy bodies (LBs). Misfolded alpha-synuclein aggregates within LBs and apha-synuclein (SYN) is the highest genetic risk factor for PD and DLB followed by the microtubule associated protein tau (MAPT) . At autopsy alpha-synuclein, hyper-phosphorylated tau (p-tau) and amyloid plaques are all detected in the brains of individuals with DLB. Therefore, the neuropathology of DLB overlaps with both PD and AD, and includes alpha-synuclein accumulation in LBs, p-tau and beta-amyloid deposition . Potential cerebrospinal fluid (CSF) biomarkers, including alpha-synuclein, dopamine metabolites homovanillic acid (HVA) and 3,4-Dihydroxyphenylacetic acid (DOPAC) , total tau and p-tau and amyloid beta peptides (Abeta 40/42) may be commonly shared in AD, PD and DLB. The core clinical features of DLB, include dementia and Parkinsonism in addition to hallucinations, cognitive fluctuations and rapid eye movement (REM) sleep behavior disorders (RBD) . L-Dopa replacement therapies and acetylcholinesterase inhibitors may partially control motor and cognitive symptoms, respectively in DLB. Selective Serotonin Re-uptake Inhibitors (SSRIs) and antipsychotics manage the behavioral but worsen motor symptoms in DLB. There is a major unmet medical need for further research into DLB to identify potential therapies for this disease and provide significant insights into the treatment of other Parkinsonian and memory disorders. A major challenge facing DLB is to develop a therapy that can halt neuronal death and alleviate cognitive, motor and behavioral symptoms. No therapeutic approach exists to alter the levels of neurotoxic proteins such as alpha-synuclein and halt DA and other neuronal death in DLB. One mechanism to degrade neurotoxic proteins is autophagy , which is a process by which the cell can degrade its own contents. There is evidence that autophagy is impaired in neurodegeneration , leading to failure of degradation of protein aggregates, including misfolded alpha-synuclein. Importantly, autophagy is exploited therapeutically in several diseases, including adult chronic myeloid leukemia (CML). Tyrosine kinase inhibitors (TKIs) induce autophagy, leading to destruction of rapidly dividing tumor cells in CML and degradation of neurotoxic proteins, including alpha-synuclein, beta-amyloid and p-tau in PD and AD models. Sun Pharma Advanced Research Company Limited (SPARC Ltd.) is developing K0706, for the treatment of adult patients with chronic phase, accelerated phase, or blast phase chronic myeloid leukemia (CML) that is resistant or intolerant to prior TKI therapy or Philadelphia positive acute lymphoblastic leukemia (Ph+ ALL) that is resistant or intolerant to prior TKI therapy; and its ability to slow down progression of PD. Using allometric scaling and an average human body weight of 70kg an oral dose of 15-30mg/kg once daily in mice corresponds to an oral human equivalent dose (HED) of 85-160 mg which is within the tolerated dose in both CML and PD. Therefore, the effects of a sachet of 192 mg powder of K0706 (equivalent to 96 mg capsule of K0706 ) and a sachet of 384 mg powder of K0706( equivalet to 192 mg capsule of K0706) and a sachet of matching placebo taken daily by mouth for 12 weeks, followed by a 4 week wash-out period will be evaluated in individuals diagnosed with DLB. The data obtained from this study will serve as a proof of concept for future placebo-controlled, double-blind studies in patients diagnosed with DLB, AD, or PD.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Capable of providing informed consent and complying with study procedures. Subjects who are unable to provide consent may use a Legally Authorized Representative (LAR)
3. Age of 25-90 years, medically stable
4. Clinical diagnosis of DLB according to McKeith et al (https://www.ncbi.nlm.nih.gov/pubmed/28592453) with both dementia MoCA≥14 and Parkinsonian defined as bradykinesia in combination with rest tremor, rigidity or both UPDRS I-III ≤ 50 and UPDRS-III between 20-40.
5. Dementia and Parkinsonism must be present with at least one other symptom such as fluctuation, visual hallucinations or REM sleep behavioral disorder (RBD)
6. Stable on Levodopa no more than 800mg daily, acetylcholinesterase inhibitors, dopamine agonists for at least 6 weeks
7. Stable on monoamine oxidase inhibitors (MOA-B) for at least 4 weeks before enrollment and during the trial
8. Stable concomitant medical and/or psychiatric illnesses in the judgement of the PI
9. Corrected QT interval (QTc) 350-470 ms, inclusive
10. Participants must be willing to undergo Lumbar puncture (LP) at baseline and 3 months after treatment.

Exclusion Criteria:

1. Medical history of liver or pancreatic disease, GI ulcers and Chron's disease, kidney, GI, or blood problems
2. Abnormal liver function defined as Aspartate aminotransferase ( AST) and/or Alanine aminotransferase (ALT) > 100% the upper limit of the normal
3. Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal or proteinuria
4. History of Human immunodeficiency virus (HIV), clinically significant chronic hepatitis, or other active infection
5. Hypokalemia, hypomagnesaemia, or long QT syndrome- QTc≥471 ms or concomitant drugs known to prolong the QTc interval and history of any cardiovascular disease, including myocardial infarction or cardiac failure, angina, arrhythmia
6. History or presence of significant cardiac conditions including: cardiovascular or cerebrovascular event (e.g. myocardial infarction, unstable angina, or stroke), congestive heart failure, first, second- or third-degree atrioventricular block, sick sinus syndrome, or other serious cardiac rhythm disturbances, any history of Torsade de Pointes.
7. Treatment with any of the following drugs at the time of screening or the preceding 30 days, and/or planned use over the course of the trial: Treatment with Class IA or III antiarrhythmic drugs (e.g. quinidine), treatment with QT prolonging drugs (www.crediblemeds.org)- excluding SSRIs (e.g. Citalopram, Escitalopram, Paroxetine, Sertraline, Duloxetine, Trazodone, etc.). Should treatment with any of these agents be required, therapy with K0706 should be interrupted.
8. Females must not be lactating, pregnant or with possible pregnancy
9. Clinical signs indicating syndromes other than DLB including, AD idiopathic PD, corticobasal degeneration, supranuclear gaze palsy, multiple system atrophy, chronic traumatic encephalopathy, signs of frontal dementia, history of stroke, head injury or encephalitis, cerebellar signs, early severe autonomic involvement, Babinski sign
10. Current evidence or history in past two years of epilepsy, focal brain lesion, head injury with loss of consciousness or Diagnostic and Statistical Manual of Mental Disorders 4th Edition ( DSM-IV) criteria for any active major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
11. Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal or other systemic disease or laboratory abnormality.
12. Active neoplastic disease, history of cancer five years prior to screening, including breast cancer (history of skin melanoma or stable prostate cancer are not exclusionary)
13. Contraindications to LP: prior lumbosacral spine surgery, severe degenerative joint disease or deformity of the spine, platelets < 100,000, use of Coumadin/warfarin, or history of a bleeding disorder.
14. Must not be on any immunosuppressant medications
15. Must not be enrolled as an active participant in another clinical study.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Evidence of treatment-emergent adverse effects (safety and tolerability) | 12 weeks
  The investigators will determine safety and tolerability by using the occurrence of adverse events (AEs) of interest, including myelosuppression, urinary, pancreatic and hepatic disorders, gastrointestinal (GI), kidney disorders, Corrected QT-interval (QTc)prolongation as per SPARC Ltd Investigator Brochure (IB).

SECONDARY OUTCOMES:
Measurement of K0706 concentration in plasma | 12 weeks
  Concentration of K0706 will be measured in the plasma
Measurement of K0706 concentration in CSF | 12 weeks
  Concentration of K0706 will be measured in the CSF
Measurement of Biomarker concentration in plasma | 12 weeks
  Concentration of DLB related plasma biomarkers, including HVA, DOPAC, Abeta40/42, total tau, ptau231/181 and total and oligomeric alpha-synuclein will be measured.
Measurement of Biomarker concentration in CSF | 12 weeks
  Concentration of DLB related CSF biomarkers, including HVA, DOPAC, Abeta40/42, total tau, ptau231/181 and total and oligomeric alpha-synuclein will be measured.

OTHER OUTCOMES:
Measurement of the effects of K0706 on Cognition using the Montreal Cognitive Assessment (MoCA) | 12 weeks
  The MoCA is designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains, including attention and concentration, executive functions, memory, language, visuo-constructional skills, conceptual thinking, calculations and orientation. Scores range between 0 and 30 where 30 is the highest score and 0 is the lowest score.
Measurement of the effects of K0706 on Cognition using the Trail Making Test (TMT) | 12 weeks
  The Trail Making Test (TMT) is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. The time to complete the test is measured.
Measuring the effects of K0706 on Cognition using the Alzheimer's Disease Assessment Scale - cognitive (ADAS-cog). | 12 weeks
  ADAS-cog aims to evaluate cognitive impairment in Alzheimer's disease. ADAS-cog was included in this LBD study to better capture potential changes in activities of daily living (ADL) and non-ADLs and severity of cognitive impairment. Points for errors in each task are added up and the greater the dysfunction, the greater the score.
Measuring the effects of K0706 on Behavior using the Alzheimer's disease Cooperative Study-Activity of Daily Living scale. | 12 weeks
  ADCS-ADL is an activity of daily living inventory to assess functional performance. Using a structured interview format, study partners are queried as to whether participants attempted each item in the inventory during the prior 4 weeks and their level of performance. The ADCS-ADL includes some items from traditional basic ADL tests as well as instrumental (complex) activities of daily living. It is a 23 item scale that provide a total score from 0-78 with a lower score indicating greater severity.
Measuring the effects of K0706 on Behavior using the Neuropsychiatric Inventory (NPI) | 12 weeks
  The NPI is a multi-item instrument to assess psychopathology in Azheimer's disease based on interview with the study partner. The NPI evaluates both the frequency and severity of 10 neuropsychiatric disturbances. Frequency assessments range from 1 (occasionally, less than once per week) to 4 (very frequently, once or more per day or continuously) as well as severity (1=mild, 2=moderate, 3=severe). The overall score and the score for each subscale are the product of severity and frequency.
Measuring the effects of K0706 on Behavior using the Clinical Assessment of Fluctuation (CAF) | 12 weeks
  The CAF consists of seven items of confusional behavior (falls, fluctuation, drowsiness, attention, disorganized thinking, altered level of consciousness, communication), scores for which are summed to provide a severity score for fluctuating confusion ranging from 0 to 21.
Measuring the effects of K0706 on Behavior using the Irritability-Apathy Scale (IAS) | 12 weeks
  The IAS measures apathy and irritability in patients with dementia. The IAS is a 28-item self-administered questionnaire collecting information about different aspects of irritability and apathy utilizing a 0-3 scale for each item to indicate severity. Both a patient and a study partner version can be administered. The IAS will be completed separately by Subjects and Study Partners. A higher total score indicates higher severity.
Measuring the effects of K0706 on Behavior using the Problem Behaviors Assessment short form (PBA-s) | 12 weeks
  PBA-s is a structured interview in which a trained interviewer rates the frequency and severity of neuropsychiatric symptoms through observation and the reporting of the Subject and Study Partner. Symptoms rated include depressed mood, suicidal ideation, anxiety, irritability, angry or aggressive behavior, apathy, perseverative thinking or behavior, obsessive-compulsive behaviors, delusional or paranoid thinking, hallucinations, and disoriented behavior. Each behavioral problem is rated for both severity and frequency on a 0-4- point scale; severity and frequency ratings are then multiplied to provide an overall score for each symptom.
Measuring the effects of K0706 on Motor Function by using the Unified Parkinson's Disease Rating Scale (UPDRS)-I-III. | 12 weeks
  UPDRS-I-III is used to follow the longitudinal course of Parkinson's disease. The UPDRS is made up of these sections: Part I: evaluation of mentation, behavior, and mood. Part II: self-evaluation of the activities of daily life (ADLs) Part III: clinician-scored monitored motor evaluation. Part IV: complications of therapy. Part V: Hoehn and Yahr staging of severity of Parkinson's disease. Part VI: Schwab and England ADL scale.
Measuring the effects of K0706 on Motor Function by using the Timed-Up-And-Go (TUG). | 12 weeks
  Timed Up and Go (TUG) is an assessment of mobility, balance, walking ability, and fall risk. It measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L Pagan, MD, Principal Investigator — Georgetown University
Locations (1):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://sites.google.com/a/georgetown.edu/moussa-lab/home3 — https://neurology.georgetown.edu/translational_neurotherapeutics